CLINICAL TRIAL: NCT03990740
Title: Myofibroblastic Transformation Secondary to Epithelial-stromal Interactions in the Keratoconus (MYKE)
Brief Title: Myofibroblastic Transformation Secondary to Epithelial-stromal Interactions in the Keratoconus
Acronym: MYKE
Status: Withdrawn | Type: Observational
Why Stopped: Logistical difficulties : protocol never finalized nor submitted
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: EGN_2017_22
Record Dates: First submitted 2019-06-11; First posted 2019-06-19 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Keratoconus
Keywords: Metalloproteinase; Glycoprotein; Cornea; Direct epithelial-stromal interactions; Fibroblasts; Myofibroblasts
MeSH Terms: conditions — Keratoconus; Corneal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients suffering from keratoconus and requiring a first optical corneal transplant
  Interventions: Procedure: Corneal sampling
- Controls: Patients with an indication of orbital exenteration operation due to an orbital tumor
  Interventions: Procedure: Corneal sampling

INTERVENTIONS:
Procedure: Corneal sampling — Corneal samples will be taken during corneal transplants for cases and orbital exenterations for controls. The mRNA (messenger ribonucleic acid) will be extracted and a retrotranscription will be made to obtain cDNA (complementary DNA). A qPCR (quantitative polymerase chain reaction) will be able to quantify the expression of alpha-SMA, MMP 1-2-3 and 9, and EMMPRIN.

SUMMARY:
Keratoconus is characterized by a thinning of the cornea, which causes a decrease in visual acuity due to astigmatism.

Publications suggest that keratoconus is linked to chronic inflammation (increase in pro-inflammatory cytokines and metalloproteinases (MMP). Direct epithelial-stromal interactions (D-ESI) have a role in the induction of metalloproteinases (MMP) and the differentiation of fibroblasts into myofibroblasts via an EMMPRIN membrane glycoprotein (extracellular matrix membran MMP inducer - CD 147). On a healthy cornea, EMMPRIN's effects are prevented by a lack of contact between epithelial and stromal cells through a basement membrane, which is altered in the keratoconus The hypothesis is that stromal thinning of the keratoconus could be related to increased expression of EMMPRIN by epithelial and stromal cells (resulting in increased MMP synthesis), with a preponderance at the most deformed areas.

The main objective is to demonstrate a transformation of fibroblasts to myofibroblasts in the corneal stroma of keratoconus patients.

ELIGIBILITY:
Inclusion Criteria:

* For the cases :

  - Suffering from keratoconus and requiring a first optical corneal transplant
* For the controls:

  * Orbital exenteration operation due to an orbital tumor
  * Absence of any anomaly of the ocular surface observed during the slit lamp examination at the last preoperative consultation

Exclusion Criteria:

* For the cases:

  * Keratoconus patient requiring a tectonic corneal transplant
  * Known pregnancy, or breastfeeding
* For the controls:

  * History of orbital radiotherapy
  * History of corneal surgery
  * History of corneal surface tumour
  * Eye surface abnormality noted in the preoperative period
  * Known keratoconus
  * Known pregnancy, or breastfeeding
  * Secondary exclusion if a keratoconus is diagnosed during the immunohistochemical analysis by visualization of Bowman membrane interruption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Keratoconus patients requiring first optical corneal transplantation and controls with indication of orbital exenteration due to an orbital tumor.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Comparison of alpha-SMA's (Smooth Muscle Actin) messenger RNA expression evaluated by quantitative PCR (RT-qPCR) in corneal stroma in keratoconus patients compared to non-keratoconus controls | 12 hours

IPD SHARING:
Plan to Share IPD: No